CLINICAL TRIAL: NCT02331251
Title: A Phase Ib/II Study of Pembrolizumab Plus Chemotherapy in Patients With Advanced Cancer (PembroPlus)
Brief Title: Study of Pembrolizumab Plus Chemotherapy in Patients With Advanced Cancer (PembroPlus)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI not longer at site.
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PembroPlus
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Advanced Cancer; Breast Cancer; Sarcoma; Pancreatic Cancer; Small Cell Lung Cancer; Ovarian
MeSH Terms: conditions — Breast Neoplasms; Sarcoma; Pancreatic Neoplasms; Small Cell Lung Carcinoma | interventions — pembrolizumab; Gemcitabine; Docetaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Vinorelbine; Irinotecan; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Gemcitabine 1000 mg/m2 on day 1 and day 8 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine
- Arm 2 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Gemcitabine 900 mg/m2 on day 1 and 8 and docetaxel 75 mg/m2 on day 8 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Docetaxel
- Arm 3 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2 on day 1 and day 8 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Arm 4 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Gemcitabine 1000 mg/m2 and vinorelbine 25 mg/m2 on day 1 and day 8 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Vinorelbine
- Arm 5 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Irinotecan 300 mg/m2 on day 1 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Irinotecan
- Arm 6 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks Liposomal doxorubicin 30 mg/m2 on day 1 every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Keytruda
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: Docetaxel
  Other Names: Taxotere
  Arms: Arm 2
Drug: Nab-paclitaxel
  Other Names: Abraxane
  Arms: Arm 3
Drug: Vinorelbine
  Other Names: Navelbine
  Arms: Arm 4
Drug: Irinotecan
  Other Names: Camptosar
  Arms: Arm 5
Drug: Liposomal Doxorubicin
  Other Names: Doxil
  Arms: Arm 6

SUMMARY:
The Phase Ib and II cohorts will enroll patients with metistatic solid tumors.

Phase II only will enroll the following patients:

Patients with metastatic sarcoma to be enrolled in the following 4 arms: pembro plus gemcitabine, pembro plus gemcitabine and docetaxel, pembro plus gemcitabine and vinorelbine, and pembro plus liposomal doxorubicin.

Patients with metastatic pancreatic adenocarcinoma to be enrolled in the pembro plus gemcitabine and nab-paclitaxel arm.

Patients with extensive-stage small cell lung cancer to be enrolled in the pembro plus irinotecan arm.

Patients with ER+ breast cancer to be enrolled in the pembro and vinorelbine arm.

Patients with ovarian cancer to be enrolled in the pembroplus liposomal doxorubicin arm.

Patients with metastatic TNBC (ER/PR/HER2 negative) to be enrolled in the pembro plus gemcitabine arm.

DETAILED DESCRIPTION:
Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient at least 18 years old and has definitive histologically or cytologically confirmed metastatic solid tumor 2. Patient has one or more metastatic tumors measurable by CT scan (or PET/CT, if patient is allergic to CT contrast media) 3. The investigator will select the appropriate treatment arm for the patient with the following requirements: (a) Patients cannot have had prior progression or intolerance on the single agent chemotherapy and then enrolled on an arm with that same single agent chemotherapy plus pembro (b) The chemotherapy on the arm selected must be considered standard of care or listed in the NCCN guidelines (www.nccn.org) for that cancer type 4. Have recovered from acute toxicities of prior treatment:

1. > 3 weeks must have elapsed since receiving any investigational agent
2. > 2 weeks must have elapsed since receiving any radiotherapy, or ≥ 3 weeks or 5 half-lives whichever is shorter for treatment with cytotoxic or biologic agents (≥ 6 weeks for mitomycin or nitrosoureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted 5. Patient has adequate biological parameters as demonstrated by the following blood counts at time of screening: 6. Absolute neutrophil count (ANC) > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 9 g/dL 7. Serum creatinine ≤2.0, total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 5 times the upper limit of normal (ULN) range (except: for the nab-paclitaxel containing arm, bilirubin ≤ 1.25 times the ULN and for the docetaxel containing arm, bilirubin must be within institutional normal limits and AST/ALT ≤ 1.5 times the ULN) 8. Thyroid stimulating hormone (TSH) within institutional normal limits. If TSH is above the upper limit of normal range, then a free T4 within institutional normal limits is acceptable 9. Persistent prior systemic therapy non-hematologic AE grade ≥ 2 (except alopecia or correctable electrolyte abnormality with supplementation) 10. Patient has a Karnofsky performance status (KPS) ≥ 70 11. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 4 months following the last dose of pembrolizumab and 30 days following the last dose of chemotherapy on this trial, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial Phase II only

   1. Patients must have metastatic sarcoma to be enrolled in the following 4 arms: pembro plus gemcitabine, pembro plus gemcitabine and docetaxel, pembro plus gemcitabine and vinorelbine, and pembro plus liposomal doxorubicin
   2. Patients must have metastatic pancreatic adenocarcinoma to be enrolled in the pembro plus gemcitabine and nab-paclitaxel arm
   3. Patients must have extensive-stage small cell lung cancer to be enrolled in the pembro plus irinotecan arm

Exclusion Criteria:

1. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
2. Serious non-healing wound, ulcer, or bone fracture
3. Patient has known brain metastases, unless previously treated and well-controlled for at least 1 month (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart)
4. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
5. Patient has known active infection with HIV, hepatitis B, or hepatitis C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol)
6. Requiring daily corticosteroid dose ≥ 10 mg prednisone or equivalent per day
7. Patient has undergone major surgery, other than diagnostic surgery (e.g., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study
8. Patient has a history of allergy or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the events outlined in the Contraindication or Special Warnings and Precautions sections of the product or comparator SmPC or Prescribing Information
9. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity
10. Patient will be receiving any other anti-cancer therapy during participation in this trial
11. Prior treatment with pembro. Receipt of other PD-1 inhibitors or PD-L1 inhibitors is allowed
12. Active or prior documented autoimmune disease requiring systemic treatment within the past 2 years Phase II portion only

1. Patients with a history of more than one primary cancer, with the exception of:

1. curatively resected nonmelanomatous skin cancer;
2. curatively treated cervical carcinoma in-situ; or
3. other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the 2 years prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Determine the recommended phase 2 dose | 3 weeks
  Objective for phase Ib: Determine the recommended phase 2 dose (RP2D) of chemotherapy in combination with pembrolizumab (pembro) in subjects with advanced cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Sangal, MD, Principal Investigator — Western Regional Medical Center
Locations (2):
- United States (2):
  - Cancer Treatment Center of America @ Western Regional Medical Center, Goodyear, Arizona
  - Western Regional Medical Center, Goodyear, Arizona

REFERENCES:
- [Derived] Weiss GJ, Blaydorn L, Beck J, Bornemann-Kolatzki K, Urnovitz H, Schutz E, Khemka V. Phase Ib/II study of gemcitabine, nab-paclitaxel, and pembrolizumab in metastatic pancreatic adenocarcinoma. Invest New Drugs. 2018 Feb;36(1):96-102. doi: 10.1007/s10637-017-0525-1. Epub 2017 Nov 8. PMID 29119276